CLINICAL TRIAL: NCT03286686
Title: Sensori-motor and Perceptual Functions of the Posterior Parietal Cortex (PPC) in Patients With Optic Ataxia (AO) and Healthy Subjects.
Brief Title: Sensori-motor and Perceptual Functions of the PPC.
Acronym: PPCfonctions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0341; 2017-A02562-51 (Other: ID-RCB)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Optic Ataxia
Keywords: optic ataxia; posterior parietal cortex functions; multisensory integration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experience 1 (Experimental)
  Interventions: Behavioral: point targets
- Experience 2 (Experimental)
  Interventions: Behavioral: point targets
- Experience 3 (Experimental)
  Interventions: Behavioral: tactile stimulation
- Experience 4 (Experimental)
  Interventions: Behavioral: visual images
- Experience 5 (Experimental)
  Interventions: Behavioral: visual images
- Experience 6 (Experimental)
  Interventions: Behavioral: visual images

INTERVENTIONS:
Behavioral: point targets — In the experiences 1 and 2, the participant needs to point different visual targets (LED) in the dark.
  Arms: Experience 1; Experience 2
Behavioral: tactile stimulation — In the experience 3, a tactile stimulation is applied to the middle finger of the 2 hands. The participant needs to indicate into a microphone when he feels the stimulation.
  Arms: Experience 3
Behavioral: visual images — Target dots or visual images are presented on a computer screen. The participant is required to point to the targets or to react as soon as possible by pressing a response button when they are detected.
  Arms: Experience 4; Experience 5; Experience 6

SUMMARY:
To produce hand's movement directed towards a target, the investigator must combine several sensory information, such as vision or proprioception. The posterior parietal cortex (PPC) is a region of the cortex involved in this multisensory integration. A lesion of the PPC cause a visuo-motor trouble called optic ataxia but these patients also have perceptual troubles.

The aim of the study is to understand the different functions of the PPC and especially how the processes of spatial coding of the sensory information influences perception and motor planning.

In this study, the investigator want to explore the sensory motor and the perceptual performance of patients with optic ataxia compared with healthy subjects, using 6 behavioral tests.

Objectify the consequences of PPC impairment (visual-motor and perceptual consequences) on patients' quality of life and autonomy.

ELIGIBILITY:
Inclusion Criteria:

All patients and healthy subjects:

* male and female, age from 18 to 75 years included
* normal vision or corrected vision
* covered by social security
* signed written informed consent

Patients:

* neurological injury in posterior parietal cortex supported by a cerebral MRI
* present optic ataxia symptoms Healthy subjects
* no known neurological injury

Exclusion Criteria:

- unable to comply with the tasks (neurological, psychiatric, sensory or motor troubles)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2031-02-22 (Estimated); Study Completion 2031-02-22 (Estimated)

PRIMARY OUTCOMES:
response error - number of pointing error | Day 0 after each stimulation
response error -measure of reaction times | Day 0 after each stimulation
response error - percentage of right responses | Day 0 after each stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Laure PISELLA, PhD, Principal Investigator — INSERM U1028 - Impact - CRNL
Locations (1):
- U1028 INSERM - CNRS UMR 5292 Equipe ImpAct, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided